CLINICAL TRIAL: NCT00246805
Title: Post Marketing Study on Heart Rate Regularization in Patients With Permanent Atrial Fibrillation
Brief Title: Heart Rate Regularization in Patients With Permanent Atrial Fibrillation Post Marketing Study
Acronym: RARE-PEARL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic BRC (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RARE-PEARL
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Results first posted 2011-09-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2010-03

CONDITIONS: Permanent Atrial Fibrillation
Keywords: Permanent atrial fibrillation; VVI(R) pacing; rate regularization

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. VRS ON (Experimental): Patients with permanent atrial fibrillation implanted with VVI(R) pacemaker Vitatron model C20 SSIR or T20 SSIR were randomized to Function Ventricular Rate Stabilization (VRS) ON or OFF.
  This arm (1) is randomized to Function Ventricular Rate Stabilization ON.
  Interventions: Device: Vitatron pacemaker C20 SSIR or T20 SSIR models
- 2. VRS OFF (No Intervention): Patients with permanent atrial fibrillation implanted with VVI(R) pacemaker Vitatron model C20 SSIR or T20 SSIR were randomized to Function Ventricular Rate Stabilization (VRS)ON or OFF.
  This arm (2) is randomized to Function Ventricular Rate Stabilization OFF.

INTERVENTIONS:
Device: Vitatron pacemaker C20 SSIR or T20 SSIR models — VRS: special function that automatically adapts pacing rate to regularize cardiac cycles
  Arms: 1. VRS ON

SUMMARY:
The purpose of this study is to monitor heart rate regularization in patients with permanent atrial fibrillation and standard indication for single chamber rate adaptive pacing VVI(R).

DETAILED DESCRIPTION:
The RARE PEARL is a multicenter prospective, randomized, double-blinded, crossover study.

Prior entering the study the patient should be informed and should give his written consent. Besides he/she should meet all selection criteria. The Investigator has to check that all selection criteria are satisfied. Then the patient undergoes pacemaker implantation, receiving a pacemaker model C20 SSIR or T20 SSIR (or later). The ventricular lead must be bipolar independently of the manufacturer.

After pacemaker implantation, a 45 days Stabilization Period is necessary to stabilize leads and drug therapy.

At the end of the stabilization period the patient is randomized to have VRS algorithm switched either ON or OFF. The 1° Study Phase ends after 2 months. Then a cross-over takes place: VRS algorithm is switched respectively OFF or ON and the 2° Study Phase is started. Also the 2° Study Phase ends after 2 months.

The randomization will be centralized: randomization lists will be generated and managed by the sponsor. Because the patients will undergo a QoL questionnaire at each crossover phase, they will have to be blinded about the status of their VRS setting. Similarly, also the co-investigators administering the QoL questionnaires have to be blinded about the status of VRS setting. Only the principal investigator knows if the VRS algorithm is ON or OFF. The principal investigator will be instructed not to inform the patient and the co-investigators administering QoL questionnaire about the setting until after the end of the study.

The co-investigator(s) responsible for QoL questionnaire should not perform the patient follow-up at 1° and 2° Study Phase, otherwise the patient is automatically excluded from the study.

After the cross-over period (2 + 2 months) a Free Therapy Phase (3° Phase) starts. Device settings and drug therapy are left to the physician's discretion.

One year after implantation a final follow-up is scheduled. The study ends and the pacemaker can be programmed according to the physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed informed consent form
* Patient with permanent atrial fibrillation, standard indication for VVI(R) pacing, and at least 1 episode of rate irregularity in the last month
* New York Heart Association (NYHA) Class I, II, III
* Patient is able to comply with follow-up times and will comply with the protocol
* > 18 years of age

Exclusion Criteria:

* Paroxysmal atrial fibrillation
* NYHA Class IV
* Left ventricular ejection fraction (LVEF) < 35
* Patients with unstable angina
* Patients who have experienced an acute myocardial infarction or received coronary artery revascularization (CABG), or coronary angioplasty (PTCA) within 3 months prior to enrolment
* Patient candidate for cardiac surgery, or coronary angioplasty (PTCA)
* Patients who experienced a cardiovascular accident (CVA) or transient ischemic attack (TIA) with permanent disability
* Life expectancy < 12 months due to other medical conditions
* Pregnancy
* The patient is enrolled in any concurrent (drug and/or device) study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Corbucci, PhD, Study Director — Vitatron Medical Italia; Eraldo Occhetta, MD, Principal Investigator — Ospedale Maggiore della Misericordia - Novara; Gianfranco Mazzocca, MD, Principal Investigator — Ospedale di Cecina (LI)
Locations (13):
- Italy (13):
  - Divisione di Cardiologia - Ospedale Civile, Livorno, LI
  - Divisione di Cardiologia - ospedale Civile, Rieti, RI
  - Divisione di Cardiologia - Ospedale Civile, Acqui Terme
  - Divisione di Cardiologia - Az. Ospedaliera Umberto I, Ancona
  - Divisione di Cardiologia - USL 8, Arezzo
  - Divisione di Cardiologia- Ospedale di Cecina, Cecina
  - Divisione di Cardiologia - Azienda USL 12 di Viareggio, Lido di Camaiore
  - Divisione Clinicizzata di Cardiologia - Az. Ospedaliera Maggiore della Carita, Novara
  - Divisione di Cardiologia - ASL 22, Novi Ligure
  - Divisione di Cardiologia - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Divisione di Cardiologia - Azienda USL 4, Prato
  - Divisione di Cardiologia - Ospedale Maria Vittoria, Torino
  - Ospedalr di Verbania, Verbania

REFERENCES:
- [Background] Proclemer A et al, Registro Italiano Pacemaker e Defibrillatori. Bollettino Periodico 2001. G Ital Aritmol Cardiostim 2002;5:5-31.
- [Background] Wittkampf FH, de Jongste MJ, Lie HI, Meijler FL. Effect of right ventricular pacing on ventricular rhythm during atrial fibrillation. J Am Coll Cardiol. 1988 Mar;11(3):539-45. doi: 10.1016/0735-1097(88)91528-8. PMID 2449483
- [Background] Lau CP, Jiang ZY, Tang MO. Efficacy of ventricular rate stabilization by right ventricular pacing during atrial fibrillation. Pacing Clin Electrophysiol. 1998 Mar;21(3):542-8. doi: 10.1111/j.1540-8159.1998.tb00096.x. PMID 9558685
- [Background] Mazzocca G, Giovannini T, Frascarelli F, Fabiani A, Burali A, Giappichini G, Bidi G, Bernabo D, Manfredini E, Corbucci G. Heart rate regularisation in patients with permanent atrial fibrillation implanted with a VVI(R) pacemaker. Europace. 2004 May;6(3):236-42. doi: 10.1016/j.eupc.2004.02.002. PMID 15121077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: enrollment period: from january 2006 till november 2008
Groups:
- VRS ON; VRS OFF: Ventricular Rate Stabilization is a programmed function of the implanted pacemaker. After the first phase (VRS ON or OFF) patients cross-over for the second phase (VRS OFF or ON)
Period: Phase 1
Arm/Group | VRS ON | VRS OFF
Started | 34 | 33
Completed | 33 | 33
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Phase 2
Arm/Group | VRS ON | VRS OFF
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VRS ON | VRS OFF | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 34 | 33 | 67
Age Continuous [Mean (Standard Deviation); unit: years] | 80 (6) | 80 (6) | 80 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 25 | 24 | 49
Region of Enrollment [Number; unit: participants]
  Italy | 34 | 33 | 67

OUTCOME MEASURES:

1. Secondary Outcome: Evaluation of Rate Irregularity Indicators and Patient's Symptoms
Time Frame: January 2009
Reporting Status: Not Posted

2. Secondary Outcome: Number of Patients That Should Undergo Atrioventricular Nodal (AVN) Ablation
Time Frame: January 2009
Reporting Status: Not Posted

3. Secondary Outcome: Number of Patients That Should Undergo Drug Therapy in Combination With Pacing to Stabilize Heart Rate
Time Frame: January 2009
Reporting Status: Not Posted

4. Secondary Outcome: Potential Discomforts of Pacing Algorithm for Heart Rate Stabilization
Time Frame: January 2009
Reporting Status: Not Posted

5. Primary Outcome: Patients Mode Preference (VRS ON, VRS OFF, NO PREFERENCE)
Description: Evaluation of patient preference concerning the programming of a specific algorithm for automatic Ventricular Rate Stabilization (VRS): Algorithm ON vs. OFF.
Time Frame: June 2009
Measure: Number; unit: participants
Arm/Group | VRS ON | VRS OFF
Number analyzed (Participants) | 66 | 66
participants
  Preference VRS ON | 32 | 32
  Preference VRS OFF | 15 | 15
  No Preference | 19 | 19
Statistical Analysis 1: Comparison: VRS ON; VRS ON vs. VRS OFF; Test type: Superiority or Other; p < 0.0001, Z-test for proportions; Proportions = 48, 95% CI 2-sided [36 to 61]

ADVERSE EVENTS:
Arm/Group | VRS ON | VRS OFF
Serious Adverse Events (participants affected / at risk) | 2/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VRS ON (N=34) | VRS OFF (N=33)
HOSPITALIZATION (Infections and infestations) | 1 (1) | 0 (0)
HOSPITALIZATION FOR HF (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
should INVESTIGATOR contemplate publishing/presenting, he shall provide copies of any abstracts, papers, or manuscripts to sponsor for review at least 30 days prior to submittal for publication or presentation. Sponsor shall limit its review to a determination of whether Confidential Information is disclosed and to check for technical correctness and shall not attempt to censor or in any way interfere with PARTICIPATING INSTITUTION's or INVESTIGATOR's presentation or conclusions